CLINICAL TRIAL: NCT00556465
Title: Study of N-Acetylcysteine for Treatment of Overt Diabetic Nephropathy
Brief Title: Efficacy of N-Acetylcysteine in Treatment of Overt Diabetic Nephropathy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3046
Record Dates: First submitted 2007-11-09; First posted 2007-11-12 (Estimated); Last update posted 2007-11-12 (Estimated); Status verified 2007-11

CONDITIONS: Diabetic Nephropathy; Chronic Kidney Disease; Diabetes Type 2
Keywords: diabetic nephropathy; proteinuria; antioxidant
MeSH Terms: conditions — Diabetic Nephropathies; Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2; Proteinuria | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A, 1,III (Experimental): in this arm patients took 1200 mg N-acetylcysteine
  Interventions: Drug: N-acetylcysteine
- B,2, III (No Intervention)

INTERVENTIONS:
Drug: N-acetylcysteine — 600 mg of effervescent N-acetylcysteine tablet twice per day for three months
  Arms: A, 1,III

SUMMARY:
Diabetic nephropathy has become the single most frequent cause of end-stage renal disease.

On a molecular level, at least five major pathways have been implicated in glucose-mediated vascular and renal damage and all of these could reflect a single hyperglycaemia-induced process of overproduction of reactive oxygen species.

Recent studies have shown that inflammation, and more specifically pro-inflammatory cytokines play a determinant role in the development of micro- vascular diabetic complications, most of the attention has been focused on the implications of TNF-α in the setting of diabetic nephropathy.

Glutathione is the most abundant low-molecular-weight thiol, and Glutathione/ glutathione disulfide is the major redox couple in animal cells.

N-acetylcysteine is effective precursors of cysteine for tissue Glutathione synthesis.

Not only does N-acetylcysteine exhibit antioxidant properties, but it may also counteract the glycation cascade through the inhibition of oxidation.

N-acetylcysteine can also reduce the apoptosis elicited by reactive oxygen species .

Indeed, N-acetylcysteine has been shown to inhibit reactive oxygen species induced mesangial apoptosis and to be able to protect cells from glucose-induced inhibition of proliferation.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients with more than 500 mg protein in 24 hours urine protein sample
* Males and post-menopausal non-lactating and non-pregnant females.
* Age greater than or equal to 30 years of age.
* Serum creatinine less than 3.0 mg/dL (265 micromoles per liter)
* Willing and able to give informed consent

Exclusion Criteria:

* Type 1 (insulin-dependent; juvenile onset) diabetes
* Patients with known non-diabetic renal disease
* Renal allograft
* Myocardial infarction, coronary artery bypass graft surgery, or percutaneous transluminal coronary angioplasty/stent within 3 months of study entry
* Cerebrovascular accident within 3 months of study entry
* New York Heart Association Functional Class III or IV
* Known allergies or intolerance to N-acetylcysteine
* Untreated urinary tract infection or other medical condition that may impact urine protein values.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-01; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Proteinuria | 3 months

SECONDARY OUTCOMES:
blood pressure,serum creatinine,GFR,c-reactive protein, | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: mohammad mahdi sagheb, MD, Study Director — shiraz university of medical science
Locations (1):
- Mohammad mahdi sagheb, Shiraz, Fars, Iran